CLINICAL TRIAL: NCT02319980
Title: The Adult Hemorrhagic Moyamoya Surgery Study
Acronym: AHMSS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Hanqiang Jiang,MD, PhD, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAHMD 2014
Record Dates: First submitted 2014-11-28; First posted 2014-12-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Moyamoya; Stroke
MeSH Terms: conditions — Moyamoya Disease; Stroke | interventions — Cerebral Revascularization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical intervention (Active Comparator): All participants in this group will be assigned to receive extracranial-intracranial arterial bypass surgery.
  Interventions: Procedure: Extracranial-intracranial bypass surgery
- Conservative management(medical management) (No Intervention): All participants in this group will be assigned to receive conservative management or medical management which involves drug therapy as considered appropriate for medical symptoms by the treating investigator.

INTERVENTIONS:
Procedure: Extracranial-intracranial bypass surgery — All participants in this group will undergo combined cerebral revascularization surgery,namely superficial temporal to middle cerebral artery bypass (STA-MCA) and encephalo-duro-myo-synangiosis(EDMS)
  Other Names: STA-MCA Bypass and EDMS
  Arms: Surgical intervention

SUMMARY:
The aim of this study is to investigate whether extracranial-intracranial(EC-IC) bypass surgery could prevent rebleeding and improve neurological function in adult moyamoya with hemorrhagic onset.

DETAILED DESCRIPTION:
About one half of adult moyamoya patients present with hemorrhagic onset.As the bleeding events are potentially fatal, it often lead to particularly poor prognosis.However, the natural history is still poorly understood.Although the rebleeding rate is known to be extremely high,no effective therapeutic method has been established based on a worldwide consensus.

The recently published Japanese Adult Moyamoya(JAM) Trial, which is the first prospective,randomized,controlled trial focused on hemorrhagic moyamoya,showed that direct bypass surgery could reduce the rebleeding rate and improve the prognosis.However,the result was statistically marginal with a small sample size and most importantly,it failed to assess the neurological function.The effect of bypass surgery on functional outcome was uncertain.

Therefore,the AHMSS study in China is designed to compare the efficacy and safety of EC-IC bypass surgery with conservative treatment in adult moyamoya patients with hemorrhagic onset by comprehensive assessment of rebleeding rate, neurological function.

ELIGIBILITY:
Inclusion Criteria:

1. Independent in activity of daily living(The modified Rankin Scale 0-2)
2. At least one month since the most recent hemorrhagic stroke
3. The neurological deficit must be stable for more than 6 weeks
4. Bleeding in ventricle,cortex,basal ganglia,thalamus and subarachnoid space confirmed by computed tomography plain scan
5. Digital substraction angiography demonstrating progressive stenosis or occlusion in the terminal portion of the internal carotid artery and/or the initial portion of the anterior or middle cerebral arteries
6. Digital substraction angiography demonstrating formation of abnormal collateral networks(moyamoya vessels) at the base of the brain,mainly in the region of thalamus and basal ganglia
7. Digital substraction angiography demonstrating the vasculopathy appeared unilaterally or bilaterally
8. Competent to give informed consent
9. Accessible and reliable for follow-up

Exclusion Criteria:

1. Other cerebrovascular diseases(such as intracranial aneurysm or brain arteriovenous malformation) probably causing intracranial hemorrhage
2. Not independent in activity of daily living(The modified Rankin Scale 3-5)
3. Moyamoya syndrome concomitant with other hereditary or autoimmune diseases(Grave's Disease,Type I Diabetes Mellitus,Type I Neurofibromatosis et al)
4. Moyamoya disease with ruptured aneurysms located in the main stem of Willis' Circle
5. Emergent evacuation of intracerebral hematoma damaging superficial temporal artery or cortical artery
6. Emergent decompressive craniotomy causing automatically developed indirect revascularization
7. Good collateral networks formed by spontaneous anastomosis between extracranial and intracranial vessels before surgery
8. Life expectancy<1 years
9. Pregnancy
10. Unstable angina or myocardial infarction with recent 6 months
11. Blood coagulation dysfunction
12. Allergic to iodine contrast agent
13. Abnormal liver function(alanine transaminase(ALT) and/or aspartate aminotransferase(AST)>3 times of normal range)
14. Serum creatinine >3mg/dl
15. Poorly controlled hypertension(systolic BP>160 mmHg,diastolic BP>100 mmHg)
16. Poor glucose control(fasting blood glucose>16.7mmol/l)
17. Concurrent participation in any other interventional clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-05; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
All strokes & death within 30 days post-surgery and ipsilateral recurrent bleeding afterwards | within 5 years of randomization
  The number of participants who suffer from all strokes & death within 30 days post-surgery and ipsilateral recurrent bleeding afterwards within 5 years of randomization

SECONDARY OUTCOMES:
All kinds of adverse events related to surgery | up to 30 days
  The number of participants who suffer from all kinds of adverse events related to surgery within 30 days
Rebleeding on the contralateral side | up to 5 years
  The number of participants who suffer from rebleeding on the contralateral side within 5 years of randomization
Transient ischemic attack on the surgically treated side | up to 5 years
  The number of participants who suffer from TIA on the surgically treated side within 5 years of randomization
The changes from baseline in modified Rankin Scale (mRS) | at 7 days, 30 days, 6 months, 12 months, 24 months, 36 months, 60 months or end of trial
  The changes from baseline in modified Rankin Scale (mRS) at 7 days, 30 days, 6 months, 12 months, 24 months，36 months，60 months or end of trial
The changes from baseline in National Institute of Health Stroke Scale (NIHSS) | at 7 days, 30 days, 6 months, 12 months, 24 months, 36 months, 60 months or end of trial
  The changes from baseline in National Institute of Health Stroke Scale (NIHSS) at 7 days, 30 days, 6 months, 12 months, 24 months，36 months，60 months or end of trial
The changes from baseline in modified Barthel Index | at 7 days, 30 days, 6 months, 12 months, 24 months, 36 months, 60 months or end of trial
  The changes from baseline in modified Barthel Index at 7 days, 30 days, 6 months, 12 months, 24 months，36 months，60 months or end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiang Gu, MD,PhD, Study Chair — Department of Neurosurgery,Huashan Hospital,Fudan University
Locations (1):
- Department of Neurosurgery,Huashan Hospital,Fudan University, Shanghai, China

REFERENCES:
- [Background] Miyamoto S, Yoshimoto T, Hashimoto N, Okada Y, Tsuji I, Tominaga T, Nakagawara J, Takahashi JC; JAM Trial Investigators. Effects of extracranial-intracranial bypass for patients with hemorrhagic moyamoya disease: results of the Japan Adult Moyamoya Trial. Stroke. 2014 May;45(5):1415-21. doi: 10.1161/STROKEAHA.113.004386. Epub 2014 Mar 25. PMID 24668203
- [Background] Derdeyn CP. Direct bypass reduces the risk of recurrent hemorrhage in moyamoya syndrome, but effect on functional outcome is less certain. Stroke. 2014 May;45(5):1245-6. doi: 10.1161/STROKEAHA.114.004994. Epub 2014 Mar 25. No abstract available. PMID 24668205
- [Background] Scott RM, Smith ER. Moyamoya disease and moyamoya syndrome. N Engl J Med. 2009 Mar 19;360(12):1226-37. doi: 10.1056/NEJMra0804622. No abstract available. PMID 19297575
- [Background] Kobayashi E, Saeki N, Oishi H, Hirai S, Yamaura A. Long-term natural history of hemorrhagic moyamoya disease in 42 patients. J Neurosurg. 2000 Dec;93(6):976-80. doi: 10.3171/jns.2000.93.6.0976. PMID 11117870